CLINICAL TRIAL: NCT05714345
Title: A Randomized, Open-Label, Phase 2 Study Evaluating Lymphodepletion With ALLO-647, Fludarabine, and Cyclophosphamide, vs. Fludarabine and Cyclophosphamide Alone, in Subjects With Relapsed/Refractory Large B-Cell Lymphoma Receiving ALLO-501A Allogeneic CAR T Cell Therapy
Brief Title: Evaluation of Lymphodepletion With ALLO-647 in Adults With R/R Large B Cell Lymphoma Receiving ALLO-501A Allogeneic CAR T Cell Therapy
Acronym: EXPAND
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early for business reasons.
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-647-201
Record Dates: First submitted 2022-12-08; First posted 2023-02-06 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Large B Cell Lymphoma
Keywords: CAR T; Cell Therapy; Allogeneic Cell Therapy; Cellular Immuno-therapy; AlloCAR T; ALLO-501A; ALLO-647; LBCL; Lymphoma; Large B-Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lymphodepletion with ALLO-647, fludarabine, and cyclophosphamide (Experimental): ALLO-501A CAR T cells infused following lymphodepletion
  Interventions: Biological: ALLO-647; Drug: Fludarabine; Drug: Cyclophosphamide; Genetic: ALLO-501A
- Lymphodepletion with fludarabine and cyclophosphamide (Experimental): ALLO-501A CAR T cells infused following lymphodepletion
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Genetic: ALLO-501A

INTERVENTIONS:
Biological: ALLO-647 — ALLO-647 is a monoclonal antibody that recognizes a CD52 antigen
  Arms: Lymphodepletion with ALLO-647, fludarabine, and cyclophosphamide
Drug: Fludarabine — Chemotherapy for lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion
Genetic: ALLO-501A — ALLO-501A is an allogeneic CAR T cell therapy targeting CD19

SUMMARY:
The purpose of the EXPAND study is to assess the safety and clinical efficacy of ALLO-647 combined with fludarabine and cyclophosphamide compared to fludarabine and cyclophosphamide alone in a lymphodepletion regimen prior to ALLO-501A CAR T therapy in adults with relapsed or refractory large B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of relapsed/refractory large B-cell lymphoma at last relapse
* Relapsed or refractory disease after at least 2 lines of chemotherapy
* ECOG performance status 0 or 1
* Absence of significant donor (product)-specific anti-HLA antibodies (DSA)
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Active central nervous system involvement by malignancy
* Autologous or allogeneic HSCT within last 6 months prior to lymphodepletion
* Hypocellular bone marrow for age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky, United States
- Universitair Ziekenhuis Brussel, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants from the United States and Europe. The informed consent date of the first participant was 01 November 2023, and the informed consent date of the last participant was 04 December 2023. The study was terminated prior to completion for business reasons, not due to safety or efficacy concerns.
Groups:
- Lymphodepletion With Fludarabine, Cyclophosphamide, and ALLO-647 (FCA): Lymphodepletion with FCA followed by treatment with ALLO-501A arm.
  Lymphodepletion:
  * Fludarabine (F) 30 mg/m^2/day intravenously (IV) on Days -5, -4, -3
  * Cyclophosphamide (C) 300 mg/m^2/ day IV on Days -5, -4, -3
  * ALLO-647 (A) 30 mg/day IV on Days -5, -4, -3
  Treatment with ALLO-501A:
  • ALLO-501A as a single IV dose of 120 × 10^6 CAR+ T cells on Day 0
- Lymphodepletion With Fludarabine, and Cyclophosphamide (FC): Lymphodepletion with FC followed by treatment with ALLO-501A arm.
  Lymphodepletion:
  * Fludarabine 30 mg/m^2/day IV, on Days -5, -4, -3
  * Cyclophosphamide 300 mg/m^2/ day IV on Days -5, -4, -3
  Treatment with ALLO-501A:
  • ALLO-501A as a single IV dose of 120 × 10^6 CAR+ T cells on Day 0
Period: Overall Study
Arm/Group | Lymphodepletion With Fludarabine, Cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion With Fludarabine, and Cyclophosphamide (FC)
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lymphodepletion With Fludarabine, Cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion With Fludarabine, and Cyclophosphamide (FC) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  Male | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  Asian | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  Native Hawaiian or Other Pacific Islander | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  Black or African American | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  White | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  More than one race | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  Unknown or Not Reported | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  Not Hispanic or Latino | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
  Unknown or Not Reported | NA — Not providing identifying information to protect participant privacy | NA — Not providing identifying information to protect participant privacy | NA
Region of Enrollment [Number; unit: Participants]
  United States | 1 | 0 | 1
  Belgium | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) of a Lymphodepletion Regimen Containing FCA vs FC Alone Per Independent Review Committee
Description: To assess the clinical efficacy of ALLO-647 (in a lymphodepletion regimen before ALLO-501A) compared to FC alone as measured by PFS and assessed by Independent Review Committee (IRC) in subjects with R/R (Relapsed / Refractory) LBCL (Large B Cell Lymphoma).
  In this study, PFS is defined as the time from randomization to disease progression, or relapse per the Lugano classification criteria (Cheson et al, 2014) as assessed by IRC or death.
Time Frame: Up to 60 months
Population: Intent-to-Treat (ITT) Analysis Set: All randomized participants. Data does not exist as assessment of efficacy per Independent Review Committee was not performed.
Measure: Median (95% Confidence Interval); unit: Participants
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall-response Rate (ORR) of a Lymphodepletion Regimen Containing FCA vs FC Per Independent Review Committee
Description: To assess the clinical efficacy of ALLO-647 as measured by ORR and assessed by Independent Review Committee (IRC) between treatment arms.
  ORR is defined as best overall response (Complete Response and Partial Response, assessed using the Lugano classification criteria 2014; Cheson , et al, 2014) by IRC at any time up through commencement of new anti-cancer therapy or withdrawal of consent.
Time Frame: Up to 60 months
Population: ITT Analysis Set: All randomized participants. Data does not exist as assessment of efficacy per Independent Review Committee was not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

3. Secondary Outcome: Event-Free-Survival (EFS) of a Lymphodepletion Regimen Containing FCA vs FC Per Independent Review Committee
Description: To assess clinical efficacy of ALLO-647 with FC (in a lymphodepletion regimen before ALLO-501A) compared to FC alone as measured by Event-Free Survival (EFS) and assessed by Independent Review Committee (IRC) in subjects with R/R LBCL.
  EFS is defined as the time from randomization to disease progression or relapse per the Lugano classification criteria 2014 as assessed by IRC, new anti-cancer therapy, or death.
Time Frame: Up to 60 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Participants
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response (DOR) of a Lymphodepletion Regimen Containing FCA vs FC Per Independent Review Committee
Description: To characterize the efficacy of ALLO-647 as measured by Duration of Response (DOR) and assessed by Independent Review Committee (IRC) between treatment arms.
  DOR is defined as time from the first observed response to disease progression or relapse (per IRC) or death.
Time Frame: Up to 60 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Participants
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS) of a Lymphodepletion Regimen Containing FCA vs FC
Description: To characterize the efficacy of ALLO-647 as measured by OS, defined as the time from randomization to death.
Time Frame: Up to 60 months, study completion, or death, whichever occurs earlier. Specifically, OS was followed for 4.5 and 10.09 months for each participant in the FCA and FC arm, respectively.
Population: ITT Analysis Set: All randomized participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 1 | 1
Months | 4.50 [4.50 to 4.50] | 10.09 [10.09 to 10.09]

6. Secondary Outcome: Duration of Response, Event-Free Survival and Progression-Free Survival of a Lymphodepletion Regimen Containing FCA vs FC Based on Response Assessment Per Investigator Review
Description: To characterize the efficacy of ALLO-647 as measured by response rate per investigator, Duration of Response (DOR), Event-Free Survival (EFS), Progression-Free Survival (PFS), assessed by investigator assessments between treatment arms.
  DOR is defined as time from the first observed response to disease progression or relapse per investigator assessment, or death.
  EFS is defined as the time from randomization to disease progression or relapse per investigator assessment per the Lugano classification criteria, new anti-cancer therapy, or death.
  PFS is defined as time from the randomization to progression or relapse per investigator assessment per the Lugano classification criteria, or death.
Time Frame: Neither participant was a responder, therefore DOR was not followed. EFS and PFS were followed from first dose of study treatment until disease progression, subsequent anticancer therapy, or death. EFS and PFS were followed for 0.99 to 1.84 months.
Population: ITT Analysis Set: All randomized participants. Duration of Response data is not applicable since there are no responders per investigator assessment.
Measure: Median (Full Range); unit: Months
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 1 | 1
Months
  Duration of Response: number analyzed (Participants) | 0 | 0
  Progression-Free Survival | 0.99 [0.99 to 0.99] | 1.84 [1.84 to 1.84]
  Event-Free Survival | 0.99 [0.99 to 0.99] | 1.84 [1.84 to 1.84]

7. Secondary Outcome: Overall Response Rate of a Lymphodepletion Regimen Containing FCA vs FC Based on Response Assessment Per Investigator Review
Description: To characterize the efficacy of ALLO-647 as measured by response rate per investigator, Overall Response Rate (ORR), and assessed by investigator assessments between treatment arms.
  ORR in FCA vs FC alone per investigator assessment at any time up through commencement of new anti-cancer therapy or withdrawal of consent.
Time Frame: Overall Response Rate was followed until disease progression or subsequent anticancer therapy, whichever occurred earlier. Specifically, ORR was followed for 0.99 to 1.84 months for each participant in the FCA and FC arm, respectively.
Population: ITT Analysis Set: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

8. Secondary Outcome: Depth and Duration of a Lymphodepletion Regimen Containing FCA vs FC
Description: To characterize the depth and duration of lymphodepletion with and without ALLO-647, as assessed by lymphocyte count.
Time Frame: From study treatment to study discontinuation, death, withdrawal of consent, or date of initiation of another anticancer therapy, whichever occurs first, for a maximum of 9 months. Only Day 28 lymphocyte counts are available for both participants.
Population: Safety-Analysis Set: All randomized participants who received at least one (partial or complete) dose of FCA/FC or ALLO-501A. Only Day 28 lymphocyte counts are available for both participants.
Measure: Mean (Full Range); unit: cells/cubic millimeter
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 1 | 1
cells/cubic millimeter | 300 [300 to 300] | 417 [417 to 417]

9. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAEs)
Description: To evaluate the overall safety profile of ALLO-647 by comparing FCA lymphodepletion with FC lymphodepletion.
Time Frame: Up to 60 months, study completion, or death, whichever occurs earlier. TEAEs were followed for 4.5 and 10.09 months for each participant in the FCA and FC arm, respectively.
Population: Safety-Analysis Set: All randomized participants who received at least one (partial or complete) dose of ALLO-647 or ALLO-501A.
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

10. Secondary Outcome: Incidence of ALLO-501A Related Treatment Emergent Adverse Events
Description: To evaluate the overall safety profile of ALLO-501A following lymphodepletion.
Time Frame: Up to 60 months, study completion, or death, whichever occurs earlier. Related TEAEs were followed for 4.5 and 10.09 months for each participant in the FCA and FC arm, respectively.
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphodepletion with fludarabine, cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion with fludarabine, and cyclophosphamide (FC)
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From participant's first dose date of any study drug up to 60 months post ALLO-647 infusion, date of death, date of study discontinuation, or the date of initiation of another anti-cancer agent, whichever occurs first; follow up of the participants ended within 11 months after ALLO-501A infusion due to death as a result of disease progression.
Description: Safety population refers to all participants who received at least one (partial or complete) dose of ALLO-501A or ALLO-647. Aggregate analysis not performed due to small sample size (N=2).
Arm/Group | Lymphodepletion With Fludarabine, Cyclophosphamide, and ALLO-647 (FCA) | Lymphodepletion With Fludarabine, and Cyclophosphamide (FC)
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphodepletion With Fludarabine, Cyclophosphamide, and ALLO-647 (FCA) (N=1) | Lymphodepletion With Fludarabine, and Cyclophosphamide (FC) (N=1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
ALLO-647-201 (EXPAND) was a Phase 2 study that was terminated prior to completion for reasons not related to safety or efficacy concerns. No analyses of the baseline, disposition, safety, primary, secondary, nor exploratory endpoints were performed due to the limited enrollment and data collected during the study. Data were listed but not summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Statistical Analysis Plan Original (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT05714345/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Statistical Analysis Plan Amendment 1 (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT05714345/Prot_SAP_001.pdf